CLINICAL TRIAL: NCT02519374
Title: Fiber Tolerability in Children
Acronym: FITIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 14.29. NRC
Record Dates: First submitted 2015-06-08; First posted 2015-08-10 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2015-07

CONDITIONS: Signs and Symptoms, Digestive
Keywords: Fiber tolerability; Children
MeSH Terms: conditions — Signs and Symptoms, Digestive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo (including Maltodextrin)
- PROMITOR® dose 1 (Active Comparator): Investigational product dose 1
  Interventions: Drug: PROMITOR® (including Maltodextrin)
- PROMITOR® dose 2 (Active Comparator): Investigational product dose 2
  Interventions: Drug: PROMITOR® (including Maltodextrin)
- PROMITOR® dose 3 (Active Comparator): Investigational product dose 3
  Interventions: Drug: PROMITOR® (including Maltodextrin)

INTERVENTIONS:
Drug: Placebo (including Maltodextrin)
  Arms: Placebo
Drug: PROMITOR® (including Maltodextrin) — Investigational product dose 1
  Arms: PROMITOR® dose 1
Drug: PROMITOR® (including Maltodextrin) — Investigational product dose 2
  Arms: PROMITOR® dose 2
Drug: PROMITOR® (including Maltodextrin) — Investigational product dose 3
  Arms: PROMITOR® dose 3

SUMMARY:
Assessment of the digestive tolerability of the PROMITOR® .

DETAILED DESCRIPTION:
The trial will be multicenter, double-blind, placebo-controlled, randomized with a 4-arm parallel-design. The subjects wil be randomized to one of the four arms, i.e. four doses of investigational product balanced in maltodextrin, given at the doses of 6, 9 or 12 g (corresponding to 4, 6, or 8 g of fibers) twice a day with the meals of the morning and of the evening versus control (maltodextrin, no fibers) over one week of intake.

The total sample size is 40 healthy children from 8 to 12 years old, male and female.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children,
* Aged between 8 and 12 years old included
* Acceptance of the taste of the product
* Having breakfast on daily basis
* Consent and/or assent received according to regulation
* Informed consent of one of the parents/guardians (for the study to be conducted in Switzerland, in respect with the Swiss regulation) or Informed consent of both parents/guardians (for the study to be conducted in France, in respect with the French regulation)
* Parents/guardians affiliated to a health insurance (only for the study to be conducted in France, in respect with the French regulation)

Exclusion Criteria:

* Specific food regimen
* Intolerability or food allergy
* Antibiotic or any medication impacting the gut transit during the 2 weeks before the study
* Chronic gastrointestinal disease
* Gastroenteritis in the 2 weeks preceding the study
* Constipation or diarrhea based on ROMEIII criteria (in average: more than 3 stools per day or less than 3 stools per week)
* Children and parents expected not to understand and perform the trial correctly (i.e.: troubles in learning and/or speaking)
* Child in a situation which, in the opinion of the principal investigator, could interfere with the optimal participation to the study or constitute a particular risk of non-compliance
* Having participated in another clinical trial for 1 month, or currently participating in a clinical trial
* Under legal protection or deprived from his rights following administrative or judicial decision (only for the study to be conducted in France, in respect with the French regulation)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Assessment of the digestive tolerability of the Investigational Product (abdominal pain) | 7 days of intake
  Using analog visual scale
Assessment of the digestive tolerability of the Investigational Product (rumbling) | 7 days of intake
  Using analog visual scale
Assessment of the digestive tolerability of the Investigational Product (bloating) | 7 days of intake
  Using analog visual scale
Assessment of the digestive tolerability of the Investigational Product (flatulence) | 7 days of intake
  Using analog visual scale
Assessment of the digestive tolerability of the Investigational Product (stools consistency & frequency) | 7 days of intake
  Using analog visual scale

CONTACTS AND LOCATIONS:
Locations (2):
- Biofortis, Saint-Herblain, France
- Metabolic Unit, Clinical Development Unit Nestec, Lausanne, Switzerland